CLINICAL TRIAL: NCT02959580
Title: Evaluation of Topical Steroids and Surgical Treatment for Idiopathic Granulomatous Mastitis
Brief Title: Medical and Surgical Treatment for Idiopathic Granulomatous Mastitis
Acronym: MSTIGM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-breast-mastitis
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Granulomatous Mastitis
Keywords: Granulomatous; Mastitis; topical steroids
MeSH Terms: conditions — Granulomatous Mastitis; Mastitis | interventions — hydrocortisone-17-butyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- medical (Experimental): Hydrocortisone butyrate cream(0.1%) was applied to the breast by the patient twice a day on alternate days until the termination of treatment.
  Interventions: Drug: Hydrocortisone Butyrate
- surgical (Active Comparator): lesion extended excision
  Interventions: Procedure: extended excision

INTERVENTIONS:
Drug: Hydrocortisone Butyrate — topical use
  Arms: medical
Procedure: extended excision — Lesion extended excision with or without a random breast dermo-glandular flap (BDGF).
  Arms: surgical

SUMMARY:
This study evaluates the clinical response rate of topical steroids in the treatment of idiopathic granulomatous mastitis in female adults. Half of the participants will receive topical steroid and the other half will receive local wide surgical excision.

DETAILED DESCRIPTION:
Idiopathic granulomatous mastitis (IGM) is a rare benign inflammatory breast disease of unknown etiology.It may present with many findings that clinically and radiologically mimic breast cancer.

Although IGM as a disease has been known for nearly four decades, the optimal treatment approach has not been established. Surgical intervention in the form of wide surgical excision was the mainstay of treatment before 1980, and is still performed depending on local expertise and preference.

Currently,surgical treatment and systemic steroid treatment are frequently employed. With the consideration of side effects of longterm systemic (oral) steroid usage, topical steroid without systemic use were assessed and showed satisfactory curative effect. But the data concerning the use of topical steroid therapy are still very limited.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Granulomatous Mastitis

Exclusion Criteria:

* Breast Carcinoma

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
clinical response rate | six months
  The clinical response is categorized into ''completely healed,'' ''inadequately healed,'' ''stable,'' ''worsened,'' or ''relapsed'' if the lesions had once healed but symptoms returned.

SECONDARY OUTCOMES:
granulomatous mastitis recurrence | two years

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Sun, master, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Breast Surgery,Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altintoprak F, Kivilcim T, Yalkin O, Uzunoglu Y, Kahyaoglu Z, Dilek ON. Topical Steroids Are Effective in the Treatment of Idiopathic Granulomatous Mastitis. World J Surg. 2015 Nov;39(11):2718-23. doi: 10.1007/s00268-015-3147-9. PMID 26148520
- [Background] Sheybani F, Naderi HR, Gharib M, Sarvghad M, Mirfeizi Z. Idiopathic granulomatous mastitis: Long-discussed but yet-to-be-known. Autoimmunity. 2016 Jun;49(4):236-9. doi: 10.3109/08916934.2016.1138221. Epub 2016 Feb 1. PMID 26829298
- [Background] Benson JR, Dumitru D. Idiopathic granulomatous mastitis: presentation, investigation and management. Future Oncol. 2016 Jun;12(11):1381-94. doi: 10.2217/fon-2015-0038. Epub 2016 Apr 12. PMID 27067146